CLINICAL TRIAL: NCT03800238
Title: Telehealth Powerful Tools for Caregivers Effectiveness Study
Acronym: TPTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University Wisconsin (Other)
Responsible Party: Principal Investigator, Katrina Serwe, Associate Professor, Concordia University Wisconsin
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ConcordiaUW
Record Dates: First submitted 2019-01-07; First posted 2019-01-11 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Caregivers
Keywords: caregiver; wellness; telehealth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data will be collected via survey and data analysis will be conducted blinded to study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Delivery Format (Experimental): This group will participate in the Powerful Tools for Caregivers program using a telehealth delivery method.
  Interventions: Behavioral: Telehealth Delivery Format
- Standard Delivery Format (Active Comparator): This group will participate in the Powerful Tools for Caregivers program in person.
  Interventions: Behavioral: Standard Delivery Format

INTERVENTIONS:
Behavioral: Telehealth Delivery Format — Participants will engage in a 6-week Powerful Tools for Caregivers program delivered via telehealth.
  Arms: Telehealth Delivery Format
Behavioral: Standard Delivery Format — Participants will engage in a 6-week Powerful Tools for Caregivers program delivered in the traditional in-person format.
  Arms: Standard Delivery Format

SUMMARY:
The purpose of this research is to examine the efficacy of telehealth as a delivery format for an education-based caregiver wellness program focusing on self-care. The study will examine two research questions. 1) Are outcomes equivalent for caregivers in an education based-wellness program delivered via telehealth and one delivered in person as measured by a general rating of health, the Center for Epidemiologic Studies Depression Scale - Revised (CESD-R), self-care behaviors (health self-care neglect, frequency of stress management and relaxation activities, and exercise frequency), self-efficacy, use of community resources, and the Bakas Caregiving Outcomes Scale (BCOS)? 2) Is class attendance equivalent for classes delivered via telehealth and in person? This research involves a specific education-based caregiver wellness program called Powerful Tools for Caregivers (PTC). PTC is an evidence-based six-week program that addresses caregiver health by promoting self-care. Collaborating community organizations offer the program at little to no cost.

This study will employ a quasi-experimental nonequivalent pretest-posttest design to compare outcomes from in-person to telehealth delivered PTC classes. PTC classes are conducted by a pair of class leaders who model concepts. Each pair of class leaders will conduct both a telehealth and in-person PTC class. Collaborating community organizations will recruit 105 caregivers to attend PTC classes delivered by 7 pairs of class leaders.

Telehealth classes will use VSee software to allow caregivers to participate in the PTC program synchronously via secure videoconferencing from their own home. VSee is a free software program designed to deliver secure telehealth services. Class leaders will guide participants in installation of the software on their home computer.

Participants will undergo assessment one week before and one week after the PTC program, and at six-month follow up. Outcome measures replicate previous PTC research and add additional outcomes meaningful to caregiver wellness. Statistical analysis will include descriptive statistics and a mixed design analysis of variance including repeated measures to examine differences in the variables of interest over time.

DETAILED DESCRIPTION:
Purpose

An estimated 43.5 million Americans serve as an unpaid caregiver over the course of a year. Caregivers are a valuable part of healthcare systems, providing a framework for the medical system to work in the home. Caregivers assist in patient follow through with medical advice, transportation to medical appointments, activation of emergency medical services, and promotion of patient quality of life. Caregivers are an asset to the healthcare system, as they reduce overall healthcare costs; in 2013, unpaid care was estimated at 470 billion dollars a year in the United States. Unfortunately, caregivers are at risk for both physical and mental health problems. In-person programs do exist that are designed to help caregivers care for themselves and mitigate their increased health risks. However, many caregivers are unable to attend such programs.

Caregivers face barriers to accessing wellness programming due to lack of time, distance from service delivery locations, availability of services, and health or caregiving demands limiting the ability to leave home. Telehealth offers a solution to many of the barriers caregivers report. Telehealth is the use of technology to deliver healthcare services at a distance. Telehealth allows people access to services regardless of physical location, availability of transportation, and availability of respite care. Telehealth also reduces travel related costs for both providers and clients. While telehealth may provide a solution to increase access to services for those who face barriers to in-person services, there is limited information on the efficacy of telehealth delivered services. No studies have been reported that directly compare outcomes from telehealth and in-person wellness programs for caregivers.

This research will fill a needed gap to inform service delivery decision making related to telehealth delivered programming for caregivers. Consequently, the overall goal of this proposed research is to determine the efficacy of translating the PTC program to a telehealth delivery format. The specific objectives are: 1) To determine whether the outcomes are different for caregivers in a PTC program delivered via telehealth compared to one delivered in person. 2) To examine program attendance and reasons for missed sessions.

These objectives will be addressed by examining the following outcomes: 1) a general rating of health, 2) the Center for Epidemiologic Studies Depression Scale - Revised (CESD-R), 3) self-care behaviors (health self-care neglect, frequency of stress management and relaxation activities, and exercise frequency), self-efficacy, use of community resources, 4) the overall caregiving experience as measured by the Bakas Caregiving Outcomes Scale (BCOS), and 5) class attendance including reasons for missed classes.

The existing program that this study proposes to examine is Powerful Tools for Caregivers, which has demonstrated positive outcomes for caregivers when delivered in-person. These benefits include reduced health risk behaviors; increased frequency in participation in self-care activities such as relaxation, exercise, and use of stress management techniques; demonstrate increased self-efficacy; lower stress levels; and report decreased caregiver burden. If the telehealth delivery method is proven effective by this research, more caregivers will be able to receive these benefits, thereby promoting positive health behaviors that prevent physical and mental health problems in this at-risk population.

PTC is an evidence-based six-week program that addresses caregiver health by promoting self-care. Collaborating community organizations offer the program at little to no cost. A preliminary feasibility study was done to prepare for the proposed research. The feasibility study involved four caregivers. Consistent class attendance and Telehealth Usability Questionnaire scores demonstrated the telehealth delivery format was feasible, and qualitative themes indicated caregivers had a positive experience. A pilot study was then conducted involving 18 caregivers in four PTC groups in four different states and examined both caregiver outcomes and the class leader experience of delivering PTC via telehealth. Results have informed the design of this proposed study.

Methodology

The proposed study is a collaboration between the National PTC Office, collaborating community agencies, and the principal investigator (PI) at Concordia University Wisconsin (CUW). The National PTC Office will provide supervision to assure fidelity to the PTC program. The National PTC Office will assist with recruiting existing PTC Class Leaders who are certified Master Trainers (those who are both certified PTC class leaders and certified to train other class leaders) to conduct PTC classes. PTC class leaders will be selected through an application process to meet criteria for experience in leading classes and to represent a diverse geographical region. These class leaders will undergo human subjects research training and work with the PI to assure compliance with the research protocol.

The proposed study will employ a quasi-experimental nonequivalent pretest-posttest design to compare outcomes from in-person to telehealth delivered PTC classes. PTC classes are conducted by a pair of class leaders who model concepts. Each pair of class leaders will conduct both a telehealth and in-person PTC class. This will control for the influence of class leader personality on outcomes.

Collaborating community organizations will recruit 105 caregivers to attend PTC classes delivered by seven pairs of class leaders. Class sizes will be unequal due to necessity. Traditional in-person PTC programs are delivered to groups of 10 caregivers. Telehealth classes are limited to five participants due to limitations in screen views and internet bandwidth. Class leaders require a video screen, as do each participant. It is distracting to view more than six video screens at once; furthermore, adding more than six participants degrades the video and audio quality due to limitations in home internet connection bandwidths. The in-person classes include partner discussions. Telehealth technology does not allow private partner discussions; however, the smaller group format is conducive to full group conversations for these aspects of the program. To control for the effect of class leaders' personality, class leaders will deliver one telehealth PTC program and one in-person PTC program. This creates unequal group sizes of 35 participants in the telehealth PTC group and 70 participants in the in-person PTC group.

The sample of 105 caregivers was determined based on a power analysis calculated using G Power software and effect sizes and attrition rates from the pilot study data. In the pilot study the CESD-R had a large effect size, while the BCOS and the other health and self-care related variables on the survey had medium to small effect sizes. The PI selected the BCOS with a Cohen's d = 0.26 for the power analysis, an alpha error probability of 0.05, and power of 0.80 to calculate sample size using G Power software. The result was a recommended sample size of 82 participants. The pilot study had a 33% rate of attrition. Planning for this level of drop out at posttest and another 33% at 6-months required an additional 15 participants be added to the sample size for a total of 97 participants in each group.

Participants will be recruited through the partnering community organizations of the PTC class leaders. Participants will be informal (unpaid) caregivers, speak English, have the cognitive ability to participate in PTC classes, and for the telehealth delivered classes have a home internet connection, computer with a camera and microphone, and demonstrate the cognitive ability to use a computer and participate in the program. PTC class leaders will screen participants to be sure they meet eligibility criteria.

Telehealth classes will use VSee software to allow caregivers to participate in the PTC program synchronously via secure videoconferencing from their own home. VSee is a free software program designed to deliver secure telehealth services. Class leaders will guide participants in installation of the software on their home computer. The telehealth process was developed and tested in earlier phases of this research.

Participants will undergo assessment one week before and one week after the PTC program, and at a six-month follow up. Outcome measures replicate previous PTC research and offer additional outcome measures meaningful to caregiver wellness. Assessments include: the Center for Epidemiologic Studies Depression Scale - Revised (CESD-R), the Bakas Caregiving Outcomes Scale (BCOS), and a PTC Taking Care of You Survey which includes items from the original PTC program outcomes research related to caregiver self-efficacy, health self-care neglect, exercise frequency, relaxation frequency, and service utilization. The survey will also include caregiver demographics and questions related to socialization. The CESD-R is an established tool to assess symptoms of depression and the BCOS captures both positive and negative aspects of the caregiver experience. Both tools have established reliability and validity. The three assessment tools will be delivered via one secure electronic survey link issued by the PI. PTC class leaders will record attendance and reasons for any missed classes.

Data Analysis

Microsoft Excel and SPSS version 25 software will be used for statistical analysis. Statistical analysis will include descriptive statistics, and a mixed design or split plot analysis of variance (ANOVA), which includes repeated measures, to examine differences in the variables of interest over time: CESD-R score, BCOS score, class attendance, caregiver self-efficacy, health self-care neglect, exercise frequency, relaxation frequency, frequency of service utilization, and frequency of socialization. Groups (telehealth delivered group n = 35 and in-person delivery model n = 70) will be analyzed for differences prior to running ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* informal (unpaid) caregivers for an adult with a chronic condition
* speak English
* cognitive ability to participate in PTC classes
* for the telehealth delivered classes have a home internet connection, computer with a camera and microphone, and demonstrate the cognitive ability to use a computer and participate in the program

Exclusion Criteria:

• non-English speaking (the PTC program and materials will be delivered in English; participants will need to be proficient in English to engage with the other members of the class)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) | Assessing change in response to participation in the Powerful Tools for Caregivers (PTC program): Baseline/ 1 week prior to participation in PTC program, 1 week after completion of the PTC program, and 6-months after completion of PTC program.
  Questionnaire assessing symptoms of depression; each question is rated on a 5-point Likert scale; total scores range from zero to 80 with a higher score indicating greater symptoms of depression.
Bakas Caregiving Outcomes Scale (BCOS) | Assessing change in response to participation in the Powerful Tools for Caregivers (PTC program): Baseline/ 1 week prior to participation in PTC program, 1 week after completion of the PTC program, and 6-months after completion of PTC program.
  Questionnaire assessing the caregiving experience (includes both positive and negative changes related to caregiver role); each question is rated on a 7-point Likert scale; total scores can range from 15 10 105 with a higher score indicating a more positive caregiving experience.
Custom created questionnaire: PTC Taking Care of You Survey | Assessing change in response to participation in the Powerful Tools for Caregivers (PTC program): Baseline/ 1 week prior to participation in PTC program, 1 week after completion of the PTC program, and 6-months after completion of PTC program.
  PTC Taking Care of You Survey which includes questions related to caregiver self-efficacy, health self-care neglect, exercise frequency, relaxation frequency, and service utilization. The survey will also include caregiver demographics and questions related to socialization.

CONTACTS AND LOCATIONS:
Overall Officials: Katrina M Serwe, PhD, Principal Investigator — Concordia University Wisconsin
Locations (13):
- United States (12):
  - OPICA Adult Day Program, Los Angeles, California
  - Health Projects Center, Santa Cruz, California
  - Tampa General Hospital, Tampa, Florida
  - Southeast Idaho Council of Governments Inc, Pocatello, Idaho
  - Iowa State University (ISU) Extension and Outreach, Webster City, Iowa
  - Michigan State University, Grand Rapids, Michigan
  - Lutheran Social Service, Moorhead, Minnesota
  - Executive Services Corps - NE, Plattsmouth, Nebraska
  - Concord Regional Visiting Nurse Association (VNA), Concord, New Hampshire
  - Kettering Health Network, Beavercreek, Ohio
  - Hope Grows and UPMC Health Plan, Pittsburgh, Pennsylvania
  - Jane Joyce, Morristown, Tennessee
- Central East Local Health Integration Network, Whitby, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Occupational Therapy Association. (2013). Telehealth [Position paper]. American Journal of Occupational Therapy, 67(6, Suppl.), S69-S90. https://doi.org/10.5014/ajot.2013.67S69
- [Background] Bakas T, Champion V, Perkins SM, Farran CJ, Williams LS. Psychometric testing of the revised 15-item Bakas Caregiving Outcomes Scale. Nurs Res. 2006 Sep-Oct;55(5):346-55. doi: 10.1097/00006199-200609000-00007. PMID 16980835
- [Background] Boise, L., Congleton, L., & Shannon, K. (2005). Empowering family caregivers: The powerful tools for caregiving program. Educational Gerontology, 31, 573-586. https://doi.org/10.1080/03601270590962523
- [Background] Burton LC, Zdaniuk B, Schulz R, Jackson S, Hirsch C. Transitions in spousal caregiving. Gerontologist. 2003 Apr;43(2):230-41. doi: 10.1093/geront/43.2.230. PMID 12677080
- [Background] Cohn ER, Brannon JA, Cason J. Resolving barriers to licensure portability for telerehabilitation professionals. Int J Telerehabil. 2011 Dec 20;3(2):31-4. doi: 10.5195/ijt.2011.6078. eCollection 2011 Fall. No abstract available. PMID 25945189
- [Background] Eaton, W. W., Smith, C., Ybarra, M., Muntaner, C., & Tien, A. (2004). Center of Epidemiologic Studies Depression Scale: Review and revision (CESD and CESD-R). In M.E. Maruish (Ed.), The use of psychological testing for treatment planning and outcomes assessment (3rd ed.) (pp. 363-377). Mahwah, NJ: Lawrence Erlbaum.
- [Background] National Alliance for Caregiving, & American Associate of Retired Persons Public Policy Institute. (2015, June). Executive summary: Caregiving in the U.S. Retrieved from http://www.caregiving.org/wp-content/uploads/2015/05/2015_CaregivingintheUS_Executive-Summary-June-4_WEB.pdf
- [Background] Reinhard, S. C., Feinberg, L. F., Choula, R. & Houser, A. (2015). Valuing the invaluable: 2015 update, undeniable progress, but big gaps remain (AARP Public Policy Institute Report). Retrieved from http://www.aarp.org/content/dam/aarp/ppi/2015/valuing-the-invaluable-2015-update-new.pdf
- [Background] Savundranayagam MY, Montgomery RJ, Kosloski K, Little TD. Impact of a psychoeducational program on three types of caregiver burden among spouses. Int J Geriatr Psychiatry. 2011 Apr;26(4):388-96. doi: 10.1002/gps.2538. PMID 20652873
- [Background] Serwe KM, Hersch GI, Pancheri K. Feasibility of Using Telehealth to Deliver the "Powerful Tools for Caregivers" Program. Int J Telerehabil. 2017 Jun 29;9(1):15-22. doi: 10.5195/ijt.2017.6214. eCollection 2017 Spring. PMID 28814991
- [Background] Serwe KM, Hersch GI, Pickens ND, Pancheri K. Caregiver Perceptions of a Telehealth Wellness Program. Am J Occup Ther. 2017 Jul/Aug;71(4):7104350010p1-7104350010p5. doi: 10.5014/ajot.2017.025619. PMID 28661387
- [Background] VSee. (2018). HIPAA and VSee video conferencing. Retrieved from https://vsee.com/hipaa/
- [Background] Won CW, Fitts SS, Favaro S, Olsen P, Phelan EA. Community-based "powerful tools" intervention enhances health of caregivers. Arch Gerontol Geriatr. 2008 Jan-Feb;46(1):89-100. doi: 10.1016/j.archger.2007.02.009. Epub 2007 Apr 27. PMID 17467080
- [Derived] Serwe KM, Walmsley AL. The effectiveness of telehealth for a caregiver wellness program. J Telemed Telecare. 2023 Aug;29(7):504-512. doi: 10.1177/1357633X21994009. Epub 2021 Jul 7. PMID 34233538